CLINICAL TRIAL: NCT00003644
Title: A Randomized Phase III Trial of IV Carboplatin (AUC 6) and Paclitaxel 175 mg/m2 Q 21 Days x 3 Courses Plus Low Dose Paclitaxel 40 mg/m2/wk Versus IV Carboplatin (AUC 6) and Paclitaxel 175 mg/m2 Q 21 Days x 3 Courses Plus Observation in Patients With Early Stage Ovarian Carcinoma
Brief Title: Carboplatin Plus Paclitaxel With or Without Continued Low-Dose Paclitaxel in Treating Patients With Early-Stage Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0175; NCI-2012-02291; SWOG-G0175
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2016-03

CONDITIONS: Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin, paclitaxel, low dose paclitaxel (Experimental): carboplatin, paclitaxel followed by low dose paclitaxel 4 weeks later
  Interventions: Drug: carboplatin; Drug: paclitaxel
- Carboplatin, paclitaxel (Active Comparator): carboplatin, paclitaxel
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether receiving combined carboplatin and paclitaxel plus continued low-dose paclitaxel is more effective than carboplatin and paclitaxel alone for early-stage ovarian cancer.

PURPOSE: This randomized phase III trial is studying carboplatin and paclitaxel alone too see how well they work compared to carboplatin and paclitaxel together with continued low-dose paclitaxel in treating patients with early-stage ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free interval and overall survival of patients with early stage ovarian epithelial cancer treated with carboplatin and paclitaxel with or without low-dose paclitaxel.
* Assess the frequency and severity of toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes. Treatment repeats every 21 days for 3 courses. Four weeks after the completion of paclitaxel and carboplatin, patients receive low-dose paclitaxel IV over 1 hour once a week for 24 weeks.
* Arm II: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes. Treatment repeats every 21 days for 3 courses. Patients then undergo observation.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study within 5.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial cancer of one of the following histologic cell types:

  * Serous adenocarcinoma
  * Malignant Brenner's tumor
  * Mucinous adenocarcinoma
  * Endometrioid
  * Adenocarcinoma
  * Clear cell adenocarcinoma
  * Undifferentiated carcinoma
  * Transitional cell
  * Mixed epithelial carcinoma
  * Adenocarcinoma - not otherwise specified
* Meets 1 of the following criteria:

  * Stage Ia or Ib, grade 3 or clear cell
  * Stage Ic or II, all grades/histologies
* Complete surgical staging
* No tumors of low malignant potential (borderline tumors)

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* Alkaline phosphatase no greater than 3 times normal
* SGOT no greater than 3 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No other invasive malignancies within the past 5 years except nonmelanoma skin cancer
* No major systemic medical illness expected to affect survival
* Body surface area no greater than 2.0

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No prior treatment for this malignancy except surgical staging
* No prior anticancer therapy that would preclude study participation

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 1998-10; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Mannel, MD, Study Chair — University of Oklahoma College of Medicine; David S. Alberts, MD, Study Chair — University of Arizona
Locations (151):
- United States (144):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Torrance Memorial Medical Center, Torrance, California
  - Colorado Gynecologic Oncology Group P.C., Aurora, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Tulane Cancer Center, Alexandria, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - OU Cancer Institute, Oklahoma City, Oklahoma
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Baptist Regional Cancer Center at Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Baptist Centers for Cancer Care, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Bon Secours Cancer Institute at St. Mary's Hospital, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Gynecologic Oncology Associates, Roanoke, Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
- Japan (7):
  - Kagoshima City Hospital, Kagoshima City, Kagoshima
  - Kobe Medical Center, Kobe
  - Shikoku Cancer Center, Matsuyama
  - National Kyushu Cancer Center, Minamiku
  - Tohoku University Graduate School of Medicine, Sendai
  - National Cancer Center Hospital, Tokyo
  - Tottori University Hospital, Tottori

REFERENCES:
- [Result] Mannel RS, Brady MF, Kohn EC, Hanjani P, Hiura M, Lee R, Degeest K, Cohn DE, Monk BJ, Michael H. A randomized phase III trial of IV carboplatin and paclitaxel x 3 courses followed by observation versus weekly maintenance low-dose paclitaxel in patients with early-stage ovarian carcinoma: a Gynecologic Oncology Group Study. Gynecol Oncol. 2011 Jul;122(1):89-94. doi: 10.1016/j.ygyno.2011.03.013. Epub 2011 May 6. PMID 21529904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG 0175 accrued 571 patients from September 1998 to December 2006.
Groups:
- Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel: Paclitaxel 175 mg/m2 IV over 3 hours, Carboplatin AUC=6 IV every 21 days x 3 cycles Followed 4 weeks later by paclitaxel 40 mg/m2 over 1 hour every week for 24 weeks
- Paclitaxel + Carboplatin Followed by Observation: Paclitaxel 175 mg/m2 IV over 3 hours, Carboplatin AUC=6 IV every 21 days x 3 cycles, followed by observation
Period: Overall Study
Arm/Group | Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel | Paclitaxel + Carboplatin Followed by Observation
Started | 289 | 282
Completed | 274 | 268
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel | Paclitaxel + Carboplatin Followed by Observation | Total
Number analyzed (Participants) | 274 | 268 | 542
Age, Customized [Count of Participants; unit: Participants]
  Less than 40 years | 22 | 21 | 43
  40-49 years | 66 | 56 | 122
  50-59 years | 88 | 98 | 186
  60-69 years | 64 | 57 | 121
  >=70 years | 34 | 36 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 268 | 542
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The percent of participants with disease recurrence within 5 years
Time Frame: Up to 5 years
Population: Eligible and treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel | Paclitaxel + Carboplatin Followed by Observation
Number analyzed (Participants) | 274 | 268
percentage of participants | 20.4 [15.9 to 25.9] | 23.2 [18.4 to 28.9]

2. Primary Outcome: Overall Survival
Description: Number of deaths during study and follow up.
Time Frame: up to 96 months
Population: All eligible and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel | Paclitaxel + Carboplatin Followed by Observation
Number analyzed (Participants) | 274 | 268
Participants | 44 | 53

3. Primary Outcome: Number of Participants With Adverse Events Grade 3 or Greater
Description: Toxicities, Grade 3 or greater (CTC version 2.0) by treatment arm for all treated participants
Time Frame: Throughout study treatment lasting up to 24 weeks
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3 & Above Toxicity Paclitaxel + Carboplatin x 24 Cycles: Paclitaxel 175 mg/m2 IV over 3 hours, Carboplatin AUC=6 IV every 21 days x 3 cycles Followed 4 weeks later by paclitaxel 40 mg/m2 over 1 hour every week for 24 weeks
- Grade 3 & Above Toxicity Paclitaxel + Carboplatin x 3 Cycles: Paclitaxel 175 mg/m2 IV over 3 hours, Carboplatin AUC=6 IV every 21 days x 3 cycles, followed by observation
Arm/Group | Grade 3 & Above Toxicity Paclitaxel + Carboplatin x 24 Cycles | Grade 3 & Above Toxicity Paclitaxel + Carboplatin x 3 Cycles
Number analyzed (Participants) | 271 | 265
Participants
  Leukopenia | 74 | 86
  Thrombocytopenia | 12 | 16
  Neutropenia | 203 | 196
  Anemia | 4 | 2
  Other hematologic | 7 | 4
  Allergy | 8 | 7
  Cardiovascular | 12 | 7
  Coagulation | 0 | 2
  Constitutional | 7 | 7
  Dermatologic | 2 | 3
  Gastrointestinal | 12 | 11
  Genitourinary/Renal | 1 | 3
  Hemorrhage | 1 | 0
  Hepatic | 1 | 1
  Infection/Fever | 15 | 11
  Metabolic | 10 | 5
  Musculoskeletal | 3 | 0
  Peripheral Neuropathy | 12 | 2
  Other Neurologic | 5 | 8
  Ocular/Visual | 1 | 0
  Pain | 15 | 12
  Pulmonary | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel | Paclitaxel + Carboplatin Followed by Observation
All-Cause Mortality (participants affected / at risk) | 44/274 | 53/268
Serious Adverse Events (participants affected / at risk) | 7/274 | 5/268
Other Adverse Events (participants affected / at risk) | 271/274 | 265/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel (N=274) | Paclitaxel + Carboplatin Followed by Observation (N=268)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 2 (3) | 0 (0)
Urinary Tract Infection With E.Coli Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Cardiac Arrythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fever with Neutropenia (Investigations) | 0 (0) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death due to Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Carboplatin Followed 4 Weeks Later by Paclitaxel (N=274) | Paclitaxel + Carboplatin Followed by Observation (N=268)
Leukopenia (Blood and lymphatic system disorders) | 247 (247) | 236 (236)
Anema (Blood and lymphatic system disorders) | 219 (219) | 209 (209)
Thrombocytopenia (Blood and lymphatic system disorders) | 122 (122) | 109 (109)
Neutropenia (Blood and lymphatic system disorders) | 255 (255) | 247 (247)
Other Hematologic (Blood and lymphatic system disorders) | 13 (13) | 13 (13)
Allergy (Immune system disorders) | 39 (39) | 24 (24)
Auditory (Ear and labyrinth disorders) | 17 (17) | 7 (7)
Cardiovascular (Cardiac disorders) | 52 (52) | 22 (22)
Coagulation (Vascular disorders) | 3 (3) | 4 (4)
Constitutional (General disorders) | 182 (182) | 159 (159)
Dermatologic (Skin and subcutaneous tissue disorders) | 215 (215) | 183 (183)
Endocrine (Endocrine disorders) | 32 (32) | 19 (19)
Gastrointestinal (Gastrointestinal disorders) | 193 (193) | 180 (180)
Hemorrhage (Vascular disorders) | 18 (18) | 11 (11)
Hepatic (Hepatobiliary disorders) | 27 (27) | 22 (22)
Infection/Fever (Infections and infestations) | 61 (61) | 25 (25)
Lymphatics (Blood and lymphatic system disorders) | 12 (12) | 3 (3)
Metabolic (Metabolism and nutrition disorders) | 53 (53) | 34 (34)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 31 (31) | 23 (23)
Neurologic (Nervous system disorders) | 73 (73) | 50 (50)
Peripheral neurologic (Nervous system disorders) | 156 (156) | 108 (108)
Ocular Visual (Eye disorders) | 27 (27) | 21 (21)
Pain (General disorders) | 164 (164) | 150 (150)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 41 (41) | 20 (20)
Sexual (Reproductive system and breast disorders) | 13 (13) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less